CLINICAL TRIAL: NCT06363539
Title: Outcome Of Treatment With Silver Nitrate Versus Topical Steroid For Umbilical Granuloma In Terms Of Healing After 3 Weeks Of Treatment
Brief Title: Silver Nitrate Versus Topical Steroid For Umbilical Granuloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children Hospital and Institute of Child Health, Lahore (Other)
Responsible Party: Principal Investigator, Muhammad Adeel Ashiq, Dr Muhammad Adeel Ashiq, Children Hospital and Institute of Child Health, Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Adeel5
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Umbilical Granuloma
Keywords: umblical granuloma; silver nitrate; topical steroid
MeSH Terms: interventions — Clobetasol; Silver Nitrate

STUDY DESIGN:
Intervention Model Description: randomized control trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- topical steroid (Experimental): topical steroid used for treatment of granuloma
  Interventions: Drug: Clobetasol Propionate .05 Mg in 100 mL TOPICAL LOTION
- silver nitrate (Experimental): silver nitrate used for umblical granuloma treatment
  Interventions: Drug: Silver Nitrate

INTERVENTIONS:
Drug: Clobetasol Propionate .05 Mg in 100 mL TOPICAL LOTION — steroid used for umblical granuloma
  Other Names: clobederm
  Arms: topical steroid
Drug: Silver Nitrate — silver nitrate used for treatment
  Other Names: silver nitrat
  Arms: silver nitrate

SUMMARY:
Umbilical granuloma is most frequent abnormality of umbilicus in infants that is defined as a moist, fleshy and pink granulation tissue at the center of umbilicus. The most commonly used treatment for umbilical granuloma is silver nitrate cauterization. Various other treatment options for umbilical granuloma include dressing with alcohol and antiseptic solutions, topical table salt, topical steroid application, suture ligation, surgical excision, electrocautery and cryotherapy. Topical steroid ointment is easily available in market, it is cheaper and safer than silver nitrate. OBJECTIVE: To compare the outcome of treatment with silver nitrate versus topical steroid for umbilical granuloma in terms of healing after 3 weeks of treatment. MATERIALS AND METHODS Study Design: Randomized Controlled Trial Setting: Department of Pediatric Surgery, Children Hospital, Lahore Duration: 6 months after approval of synopsis [Sept 20, 2022 till March 20, 2023] DATA COLLECTION PROCEDURE 2 After approval of study from hospital Ethical committee & CPSP, all patients fulfilling the inclusion criteria were admitted through the pediatric surgery outpatient department of The Children's Hospital Lahore. 354 Patients were divided in two equal groups randomly, using lottery method Group A (control group) in which silver nitrate was applied to the lesion once a week and Group B (experimental group) in which topical steroid ointment was applied to the lesion twice a day. Patients were followed after 3 weeks to see healing of umbilical granuloma. Photographs were taken before start of treatment and on regular intervals at each follow up visit. All data was collected by myself.

DETAILED DESCRIPTION:
Umbilical granuloma is most frequent abnormality of umbilicus in infants with prevalence of 1 in 500 newborns.1 Umbilical granuloma is defined as a moist, fleshy and pink granulation tissue at the center of umbilicus.2,3 Many congenital conditions such as patent urachus and persistent vitellointestinal duct can mimic umbilical granuloma but they present with discharge of urine or feces having different smell from the umbilicus.4 Characteristically the granulomas become apparent after separation of umbilical cord. Once umbilical cord is clamped during delivery, a rapid separation begins and cord spontaneously detaches within7 to15 days and disappears by 2 to 3 weeks.1,5,6 Umbilical granuloma predominantly consists of fibroblasts, copious blood vessels, endothelial and inflammatory cells in an edematous stroma with no neural elements.3,7,8 Delayed cord separation i.e. persisting cord beyond 2 - 3 weeks, occurs in the presence of an ongoing subclinical or mild infection in umbilical stump, leading to granuloma formation.7,9 Most common symptoms of umbilical granuloma are small swelling and discharge. Physical examination shows a small 1 to 10mm, soft, friable, non-tender and pale pink lesion at base of umbilicus.10,11 It can be diagnosed easily with careful history, physical examination of umbilicus 5 and type of discharge and frequently requires no further investigation. If there is any doubt about diagnosis then other diagnostic modalities can be used such as, ultrasound abdomen, contrast studies and excisional biopsy can be used to rule out other anomalies of umbilicus including urachal anomalies, vitelline duct anomalies and benign soft tissue tumors of umbilicus.6,12-15 The most commonly used treatment for umbilical granuloma is silver nitrate cauterization. 4,12 Chemical burns to the periumbilical area, eyelids and pigmentation changes are reported complications of silver nitrate cauterization. Therefore clinic application of silver nitrate is advised on outdoor basis by trained health professionals.16-18 Various other treatment options for umbilical granuloma include dressing with alcohol and antiseptic solutions, topical table salt, topical steroid application, suture ligation, surgical excision, electrocautery and cryotherapy.5,12,15,19 Topical steroid ointment for the treatment of umbilical granuloma has gained wide attention due to its advantages of effectiveness and simplicity.20,21Topical steroid exerts anti-inflammatory effects and reduce the number of fibroblasts so its beneficial for treating umbilical granuloma.8,22 Topical steroids can be applied at home by parents requiring no supervision of health care professionals. However, prolonged 6 application of topical steroid can lead to skin infections, hypopigmentation, atrophy and Cushing syndrome so long term use should be avoided.4 In a study the healing rate after 3 weeks of treatment with topical steroid ointment were almost identical to that silver nitrate cauterization as 90.4% versus 91% with no major complication.23 Another study shows; The healing rate at 3 weeks after treatment with silver nitrate and clobetasol propionate 0.05%(steroid) were compatible as 96.6% and 90% respectively with mild side effects of skin pigmentation and atrophy.21 Although multiple studies are conducted to assess the efficacy of silver nitrate cauterization but limited study is available to compare the efficacy of topical steroid treatment for umbilical granuloma. My study may help to assess the efficacy of topical steroid ointment in the treatment of umbilical granuloma. Topical steroid ointment is easily available in market, it is cheaper and safer than silver nitrate. It may help to assure the parental satisfaction as they can apply it at home safely and may reduce the burden on hospital, moreover, no similar study has been conducted in our hospital yet, and thus it may be add to the limited clinical data available and improves patient care.

ELIGIBILITY:
Inclusion Criteria:

* Umbilical granuloma as per operational definition 2. Age below 1year 3. Both male and female genders

Exclusion Criteria:

* 1.Prior treatment of umbilical granuloma either medical or surgical. 2. Umbilical anomalies as vitelline duct anomalies, urachal anomalies, soft benign tumors of umbilicus 3. Syndromic Child with any other co-morbid condition.

Ages: 1 Month to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 354 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
healing | 3 weeks
  rate of healing observed

CONTACTS AND LOCATIONS:
Overall Officials: Adeel A Gujjar, M.S, Principal Investigator — Dr Adeel Gujjar MBBS MS
Locations (1):
- Children Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
no plan of sharing